CLINICAL TRIAL: NCT05229952
Title: Assessment of Endogenous Oxalate Synthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Sonia Fargue, Assistant Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: IRB151020005-OXI
Record Dates: First submitted 2022-01-27; First posted 2022-02-08 (Actual); Results first posted 2024-12-11 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Healthy; Kidney Stone; Obesity
Keywords: Oxalate; Kidney stones; Urolithiasis; Nephrolithiasis; Urologic disease; Oxalate metabolism
MeSH Terms: conditions — Kidney Calculi; Obesity; Urolithiasis; Nephrolithiasis; Urologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Constant infusion of 13C2-oxalate (Experimental): Subjects who have passed screening, will consume a low-oxalate, normal calcium controlled diet for 5 days total. On Days 3 and 4, subjects will collect two 24-hour urines. On Day 5, they will receive a carbon 13 oxalate infusion which will occur at a constant rate for 6 hours, in the fasted state, following a priming dose. Hourly urine and twice hourly blood samples will be collected during the 6 hours. Meals will be resumed at the end of the infusion and timed urine collections will take place at home until the next day. A DXA scan will be performed to assess body composition at another date.
  Interventions: Dietary Supplement: Low-oxalate controlled diet; Other: Primed, continuous intravenous infusion of 13C2-oxalate

INTERVENTIONS:
Dietary Supplement: Low-oxalate controlled diet — Participants will consume a diet that is controlled in its contents of protein, carbohydrates, fat, calcium, oxalate, vitamin C and sodium for 5 days. Participants will be asked not to take any dietary supplements, exercise strenuously, or consume food or drink that is not provided to them.
Other: Primed, continuous intravenous infusion of 13C2-oxalate — Participants will receive a continuous intravenous administration of carbon-13 oxalate, a naturally occurring form of oxalate, over the course of several hours until steady-state is achieved, using an IV catheter, while remaining fasting.

SUMMARY:
This study aims to determine the daily rate of endogenous synthesis of oxalate using carbon 13 oxalate isotope tracer technique and a low-oxalate controlled diet.

DETAILED DESCRIPTION:
Urinary oxalate excretion is derived from both dietary sources and endogenous synthesis. This study will use low-oxalate controlled diet and intravenous infusion of the isotope tracer carbon 13 oxalate, timed with blood and urine collections, to determine the daily rate of endogenous oxalate synthesis in non-stone forming volunteers and in subjects with calcium oxalate kidney stones. A DXA scan will be used to assess body composition.

ELIGIBILITY:
Inclusion Criteria:

* Mentally competent adults, able to read and comprehend the consent form
* Body Mass Index (BMI) between 18.5 and 50 kg/m2
* Acceptable 24 hour urine collections (judged on screening)
* good health as judged from a medical history, reported medications, and a complete blood metabolic profile
* with or without history of calcium oxalate kidney stones

Exclusion Criteria:

* History of any hepatic, bowel, or endocrine disease or other condition that may influence the absorption, transport or urine excretion of ions
* Abnormal urine chemistries or blood metabolic profiles
* Poor 24 hour urine collections completed during screening, judged by 24 hour urine creatinine excretion (indicative of not collecting all urine in the 24 hour period)
* Pregnancy, intention to become pregnant in the near future, or lactation
* Aged lower than 18 or greater than 75 years
* BMI lower than18.5 or greater than 50 kg/m2

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2024-09-09 (Actual); Study Completion 2024-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Fargue, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fargue S, Wood KD, Crivelli JJ, Assimos DG, Oster RA, Knight J. Endogenous Oxalate Synthesis and Urinary Oxalate Excretion. J Am Soc Nephrol. 2023 Sep 1;34(9):1505-1507. doi: 10.1681/ASN.0000000000000176. Epub 2023 Jun 14. No abstract available. PMID 37312251

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Constant Infusion of 13C2-oxalate
Started | 23
Completed | 23
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: individuals with and without history of calcium oxalate kidney stones
Arm/Group | Constant Infusion of 13C2-oxalate
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 23
Body mass index [Mean (Standard Deviation); unit: kg/m2] | 31 (6)

OUTCOME MEASURES:

1. Primary Outcome: Endogenous Oxalate Synthesis Rate
Description: Daily oxalate synthesis rate (mg/day) determined by the 13c2-oxalate infusion method
Time Frame: day 5
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | Constant Infusion of 13C2-oxalate
Number analyzed (Participants) | 23
mg/day | 17 (4)

2. Secondary Outcome: Urinary Oxalate Excretion
Description: 24-hr urinary oxalate excretion (mg/day) after equilibration on the low-oxalate controlled diet, measured by ion chromatography coupled with mass spectrometry.
Time Frame: day 3-4
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | Constant Infusion of 13C2-oxalate
Number analyzed (Participants) | 23
mg/day | 20 (4)

3. Secondary Outcome: Urinary Creatinine Excretion
Description: 24-hr urinary creatinine excretion (g/day) after equilibration on the low-oxalate controlled diet.
Time Frame: day 3-4
Measure: Mean (Standard Deviation); unit: g/day
Arm/Group | Constant Infusion of 13C2-oxalate
Number analyzed (Participants) | 23
g/day | 1.6 (0.5)

ADVERSE EVENTS:
Time Frame: 5 days
Arm/Group | Constant Infusion of 13C2-oxalate
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-12-08): https://cdn.clinicaltrials.gov/large-docs/52/NCT05229952/Prot_SAP_000.pdf
  • Informed Consent Form (2021-03-24): https://cdn.clinicaltrials.gov/large-docs/52/NCT05229952/ICF_001.pdf